CLINICAL TRIAL: NCT05628948
Title: Vascular Lab Resource (VLR) Biorepository Study
Brief Title: Vascular Lab Resource (VLR) Biorepository
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Scott Cameron, MD, PhD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 19-1451
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases; Metabolic Disease; Peripheral Artery Disease; Carotid Disease; Aneurysmal Disease; Venous Disease; Thrombosis; Lymphedema; Lipedema; Non-Atherosclerotic Chronic Arterial Occlusive Disease; Vasculitis; Fibromuscular Dysplasia; Arterial Dissection; May-Thurner Syndrome; Thoracic Outlet Syndrome; Vasospasm
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases; Peripheral Arterial Disease; Thrombosis; Lymphedema; Lipedema; Vasculitis; Fibromuscular Dysplasia; Dissection, Blood Vessel; May-Thurner Syndrome; Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic testing such including messenger RNA sequencing (mRNA-seq), DNA sequencing including whole exome sequencing and whole genome sequencing, and protein analysis may be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study of biomarkers obtained from prospectively collected subject samples and their correlation with cardiovascular and metabolic diseases. The purpose of this initiative is to develop an enduring tool to allow for collaborative research between clinicians at Cleveland Clinic Main Campus and basic scientists at the Lerner Research Institute. This collaboration will allow resources to be available to clinical and basic researchers alike. This tool will enable research of vascular disease in the Vascular Lab and will leverage this valuable asset to the fullest extent to allow for interdepartmental collaboration.

DETAILED DESCRIPTION:
We are proposing a study of biomarkers obtained from prospectively collected subject samples and their correlation with cardiovascular and metabolic diseases. The purpose of this initiative is to develop an enduring tool to allow for collaborative research between clinicians at Cleveland Clinic Main Campus and basic scientists at the Lerner Research Institute. This collaboration will allow resources to be available to clinical and basic researchers alike. This tool will enable research of vascular disease in the Vascular Lab and will leverage this valuable asset to the fullest extent to allow for interdepartmental collaboration.

The care of subjects with vascular and metabolic diseases is very fragmentary, and they remain underserved clinically and under-studied. We will capitalize on the highly collaborative clinical environment in HVI and other clinical institutes to develop and constantly utilize a vascular biobank.

This protocol will study blood, urine, and/or stool samples and clinical data from subjects with cardiovascular and/or metabolic diseases including: peripheral artery disease, carotid disease, aneurysmal disease, chronic venous disease, thrombosis, lymphedema and lipedema, non-atherosclerotic arterial stenosis (vasculitis, fibromuscular dysplasia, arterial dissection and aneurysmal disease, May-Thurner Syndrome etc.), compressive and spastic disorders (thoracic outlet syndrome, vasospasm). This initiative will allow for the opportunity to explore pathways of thrombosis, inflammation, gut microbiome, alterations in cell signaling, lipid metabolism and other metabolic pathways in vascular diseases. Further, this study will enhance and expand ongoing efforts in the Vascular Lab to collect data for the purpose of quality control and safety. The specimen sample collection will enable biochemical and genetic testing on participants once sufficient numbers are attained.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Subjects capable of providing informed consent document
3. Subjects with diagnosed with or at risk for cardiovascular and metabolic diseases

Exclusion Criteria:

1. Known life expectancy of ≤ 6 months at the time of enrollment
2. Known current pregnancy
3. Severe Anemia (last documented hemoglobin < 7.0 g/dL)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are with or at risk for cardiovascular or metabolic disease.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
To collect blood, urine, and/or stool samples for biorepository | 10 years
  To explore pathways of thrombosis, inflammation, gut microbiome, alterations in cell signaling, lipid metabolism and other metabolic pathways in vascular diseases

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cameron, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No